CLINICAL TRIAL: NCT07323667
Title: REVIVE Zug: Impact of a Cantonal First Repsonder System on ROSC Rates and Incidence of Shockable Rhythms in Out-of-hospital Cardiac Arrest
Brief Title: A Study on the Impact of a New Canton-Wide First Responder System in Zug, Switzerland, on Survival After Adult Cardiac Arrest-Examining Early Life-Saving Organized Help, Fast Defibrillation, and Improved Outcomes for Out of Hospital Cardiac Arrest
Acronym: REVIVE Zug
Status: Enrolling by invitation | Type: Observational
Sponsor: Felix Brinkmann (Other Government)
Responsible Party: Sponsor-Investigator, Felix Brinkmann, Principal Investigator, Rettungsdienst Zug
Organization: Rettungsdienst Zug (Other Government)
Other Study IDs: 2025-01169
Record Dates: First submitted 2025-06-25; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Arrest (CA); Cardiac Arrest With Successful Resuscitation; Resuscitation; Emergency Medical Services; First Aid; Defibrillators; Cardiopulmonary Resuscitation (CPR); Bystander Effect; Survival Rate; Critical Care Medicine; Paramedical Professionals
Keywords: OHCA; Resuscitation; First responder; AED; Automated external Defibrillator; Return of spontaneous circulation; ROSC; Critical care paramedic; Emergency physician; Prehsopital care; Paramedic-led care; Physician-led care; Switzerland
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients with OHCA before the implementation of First Responder system (retropersp.): Cohort 1: Pre-Implementation Group Patients who experienced out-of-hospital cardiac arrest (OHCA) in the canton of Zug before the introduction of the comprehensive First Responder system (retrospective cohort).
- Cohort 1: Patients with OHCA after the implementation of First Responder system (propersp.): Cohort 2: Post-Implementation Group Patients who experienced out-of-hospital cardiac arrest (OHCA) in the canton of Zug after the introduction of the comprehensive First Responder system (prospective cohort).

SUMMARY:
REVIVE Zug: Improving Emergency Response for Out-of-Hospital Cardiac Arrest

Out-of-hospital cardiac arrest (OHCA) represents one of the most time-critical medical emergencies, where rapid recognition and immediate intervention are decisive for survival and neurological outcome. Early activation of emergency services, prompt initiation of cardiopulmonary resuscitation, and rapid defibrillation using automated external defibrillators (AEDs) are key components of the chain of survival. In many regions, organized First Responder systems-such as fire services, police forces, and trained lay responders supported by dispatcher-assisted instructions-arrive at the scene before emergency medical services (EMS) and initiate life-saving measures.

Evidence from multiple EMS systems indicates that the early involvement of First Responders is associated with higher rates of return of spontaneous circulation (ROSC) and improved survival to hospital discharge with favorable neurological outcomes. Regions with well-established First Responder networks consistently report better OHCA outcomes compared with regions without such systems.

In the canton of Zug, a comprehensive First Responder system has recently been implemented alongside an established hybrid EMS response model. In this system, resuscitation efforts are led either by an Emergency Physician (EP) or by a highly trained Critical Care Paramedic (CCP), depending on operational availability. Both roles operate within clearly defined competencies and provide the full scope of advanced prehospital care. This hybrid leadership model offers a unique opportunity to examine whether the professional background of the team leader influences resuscitation outcomes in real-world clinical practice.

The REVIVE Zug study aims to evaluate the impact of the canton-wide First Responder system on outcomes following OHCA. Key outcomes of interest include ROSC rates, hospital admission after cardiac arrest, the occurrence of shockable rhythms at EMS arrival, and outcomes achieved before EMS arrival. In addition, the study explores whether team leadership by an EP or a CCP is associated with differences in resuscitation outcomes. Further analyses focus on time intervals within the chain of survival, such as time from cardiac arrest to arrival of organized help and time to first defibrillation, as well as on event timing and basic demographic characteristics.

The study is based on anonymized data from established EMS quality registries and the national Swiss Reca database. By comparing OHCA cases before and after implementation of the comprehensive First Responder system, the project seeks to provide robust, practice-oriented evidence to inform future development of prehospital emergency care systems in Switzerland and comparable settings.

DETAILED DESCRIPTION:
Background and Rationale

Out-of-hospital cardiac arrest (OHCA) remains one of the leading causes of prehospital mortality and represents a medical emergency with extreme time sensitivity. Survival and neurological outcome are strongly dependent on early recognition, rapid activation of the emergency response system, immediate high-quality cardiopulmonary resuscitation, and timely defibrillation. Delays at any stage of the chain of survival substantially reduce the likelihood of return of spontaneous circulation (ROSC) and survival to hospital discharge.

Organized First Responder systems, including fire services, police units, and trained lay responders supported by dispatcher-assisted cardiopulmonary resuscitation, have been shown to strengthen the early phases of OHCA management. These responders frequently arrive before emergency medical services (EMS) and initiate life-saving interventions during the critical first minutes after collapse. Regions with structured First Responder programs consistently report higher ROSC rates, shorter time to first defibrillation, and improved survival compared with regions without such systems.

In the canton of Zug, Switzerland, EMS operates within a hybrid response model in which resuscitation teams are led either by an Emergency Physician (EP) or by a highly trained Critical Care Paramedic (CCP), depending on operational availability. CCPs have completed advanced postgraduate training and operate with a high degree of autonomy within clearly defined delegated competencies. Both EPs and CCPs are authorized to provide the full range of advanced prehospital resuscitation care. This model reflects a pragmatic approach to maintaining high-quality emergency coverage while allowing flexibility in staffing.

The coexistence of a canton-wide First Responder system and a hybrid EMS leadership model provides a unique opportunity to evaluate system-level effects on OHCA outcomes within a real-world Swiss setting. While international literature suggests that overall survival outcomes are broadly comparable between physician-led and paramedic-led resuscitations, ongoing debate persists regarding potential differences in specific subgroups or early resuscitation endpoints. At the same time, evidence increasingly emphasizes that early intervention by First Responders may have a greater population-level impact than the professional background of the advanced life support team leader.

Despite the widespread implementation of First Responder programs in Switzerland, systematic evaluation in the German-speaking regions remains limited. REVIVE Zug addresses this gap by providing a comprehensive analysis of OHCA outcomes before and after implementation of a full-coverage First Responder system, while accounting for the potential influence of EMS team leadership.

Objectives

The primary objective of the REVIVE Zug study is to assess the impact of a canton-wide First Responder system on outcomes following out-of-hospital cardiac arrest.

Primary outcomes include:

Rates of return of spontaneous circulation

Rates of hospital admission following OHCA

Occurrence of shockable cardiac rhythms at EMS arrival

Achievement of ROSC prior to arrival of EMS

Secondary objectives focus on evaluating whether the type of EMS team leadership-Emergency Physician versus Critical Care Paramedic-is associated with differences in resuscitation outcomes once EMS-led care has begun. Additional analyses examine key time intervals within the chain of survival, including time from cardiac arrest to arrival of organized help and time to first defibrillation. Event timing characteristics (such as time of day and weekday versus weekend occurrence) and basic demographic factors are also assessed to support contextual interpretation of results.

Study Design

REVIVE Zug is an ambispective observational data analysis combining retrospective and prospective cohorts. The retrospective cohort includes OHCA cases occurring prior to implementation of the comprehensive First Responder system, while the prospective cohort includes cases managed after full system deployment.

The study uses encrypted, non-genetic, health-related personal data derived from established registries, including the local EMS quality registry and the national Swiss Reca resuscitation registry. Data collection follows standardized documentation procedures using routine EMS records and case report forms. For prospective data, an additional structured case report form for First Responder interventions has been introduced to address potential documentation gaps.

Only adult OHCA cases occurring within the canton of Zug are included. Pediatric cases are excluded due to low case numbers. Cases with a documented refusal for data use are excluded.

Data Management and Statistical Approach

All data are pseudonymized at the point of entry and fully anonymized for analysis. Linkage keys are stored separately and accessible only to a limited number of specifically authorized individuals. Data are stored on encrypted, password-protected servers within the Health Directorate of the canton of Zug.

Statistical analyses are exploratory and descriptive in nature. Continuous variables are summarized using mean and standard deviation or median and range, depending on data distribution. Categorical and ordinal variables are reported as counts and proportions. Group comparisons are conducted using appropriate statistical tests based on data characteristics, including parametric and non-parametric methods. Correlation analyses are performed using established statistical coefficients as appropriate. Standard statistical software packages are used for analysis and graphical presentation.

Based on historical data, the expected annual number of OHCA cases in the study region is approximately 40 cases per year, resulting in an estimated total sample size of around 250 cases across the full study period.

Data Sources and Security

Study data originate from the Swiss Reca registry and the internal EMS quality registry, both of which have long-standing experience with standardized, pseudonymized data collection. EMS mission reports and routine documentation are archived in accordance with cantonal quality assurance procedures.

All study data are centrally stored within the Health Directorate of Zug. Access is strictly limited to authorized personnel through role-based permissions. Audit trails, access logging, and data integrity controls are in place. Data handling follows established clean-desk and information security policies.

Ethical Considerations and Regulatory Compliance

Due to the acute nature of OHCA and the high associated mortality, it is often not feasible to obtain individual informed consent retrospectively. The study therefore operates under an exemption in accordance with Article 34 of the Swiss Human Research Act for the use of anonymized health-related data. This exemption has been granted by the responsible ethics committee for Northwest and Central Switzerland.

No data are included if a written or verbal refusal has been documented. All individuals with access to coded or operational data are subject to Swiss medical confidentiality obligations and official secrecy requirements. Patient data are retained for a minimum of five years in accordance with Swiss quality assurance and regulatory standards.

The study complies with the Swiss Human Research Act and Human Research Ordinance. Any protocol amendments or changes in project responsibility are documented and reported in accordance with regulatory requirements.

Anticipated Outcomes and Relevance

REVIVE Zug aims to provide a differentiated, practice-oriented assessment of how a comprehensive First Responder system influences OHCA outcomes within a real-world EMS environment. By integrating operational data with standardized registry information, the study seeks to generate findings that are relevant to EMS system design, responder training, and emergency planning.

The results are expected to support evidence-based decisions regarding early response strategies and the organization of prehospital care. Findings will be disseminated through scientific publication and professional exchange, with the goal of informing future improvements in OHCA management in Switzerland and comparable healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older) who experienced out-of-hospital cardiac arrest (OHCA) in the canton of Zug.

Exclusion Criteria:

* Patients younger than 18 years (pediatric cases).
* Patients with a documented refusal (written or verbal) to use data for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals who experienced out-of-hospital cardiac arrest (OHCA) within the canton of Zug, Switzerland. Participants will be identified based on entries in local emergency medical services (EMS) registries and the national Swiss Reca registry. The population reflects all eligible OHCA cases attended by the Zug EMS, including both pre- and post-implementation periods of the First Responder system.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Return of Spontaneous Circulation (ROSC) prior to arrival of EMS. | Time Frame: From cardiac arrest onset (as recorded by bystander/witness or dispatch log) until EMS arrival on scene (time-stamped in EMS run sheet); assessed up to 60 minutes.
  Definition: Number and proportion of out-of-hospital cardiac arrest (OHCA) patients achieving ROSC prior to arrival of EMS.
Hospital admission after OHCA | From cardiac arrest onset until documented handover at the ED or ICU (time-stamped in EMS/hospital record); assessed up to 24 hours.
  Definition: Number and proportion of OHCA patients who are admitted to the hospital (survived to hand-over at the emergency department or ICU).
Occurrence of shockable rhythm at EMS arrival | Baseline (initial rhythm documented at EMS arrival on scene).
  Definition: Number and proportion of patients presenting with a shockable cardiac rhythm (ventricular fibrillation/pulseless ventricular tachycardia) upon first EMS assessment.

SECONDARY OUTCOMES:
Prehospital resuscitation outcome by EMS team leadership (Emergency Physician vs Critical Care Paramedic) | From EMS arrival on scene until hospital handover (ED/ICU) while in ROSC or death pronounced on scene; assessed up to 6 hours.
  Number and proportion of out-of-hospital cardiac arrest (OHCA) patients with the following prehospital resuscitation outcomes, analyzed by EMS team leadership type:
  ROSC at hospital handover: sustained return of spontaneous circulation with transport and handover at the emergency department (ED) or ICU while in ROSC, or Death pronounced on scene: termination of resuscitation with death pronounced on scene.
  Leadership category determined by EMS team leader profession (Emergency Physician [EP] or Critical Care Paramedic [CCP]) at the incident.
Time from Cardiac Arrest to Arrival of Organized Help | Baseline (index OHCA event; prehospital interval, measured once).
  Definition: Measured interval (minutes) from estimated time of OHCA to arrival of the first organized responder (EMS or First Responder).
Time to First Defibrillation | From estimated cardiac arrest onset (witness/dispatch record) until first defibrillation (defibrillator time-stamp/EMS record); assessed up to 60 minutes.
  Definition: Interval (minutes) from time of cardiac arrest to delivery of first defibrillation.
Event Timing | At cardiac arrest onset (baseline).
  Distribution of out-of-hospital cardiac arrest events by time of day (day vs. night).
Demographics (Age, Gender) | Baseline (at cardiac arrest onset)
  Descriptive analysis of patient demographics, including age and sex.
Day of week of cardiac arrest occurrence | At cardiac arrest onset (baseline)
  Distribution of out-of-hospital cardiac arrest events by weekday versus weekend.
Date and calendar distribution of cardiac arrest events | At cardiac arrest onset (baseline)
  Distribution of out-of-hospital cardiac arrest events by calendar date.

CONTACTS AND LOCATIONS:
Locations (1):
- Rettungsdienst des Kantons Zug // Emergency Medical Service of the Canton Zug, Zug, Canton of Zug, Switzerland

IPD SHARING:
Plan to Share IPD: No
At this time, we do not plan to share individual participant data (IPD) outside the study team due to data protection requirements and restrictions in the consent and ethics approval. Data may be available upon reasonable request to the corresponding author and subject to additional ethical approval. Ethic committee permission and strict Swiss data protection guidelines apply.

REFERENCES:
- [Background] Bjornsson HM, Bjornsdottir GG, Olafsdottir H, Mogensen BA, Mogensen B, Thorgeirsson G. Effect of replacing ambulance physicians with paramedics on outcome of resuscitation for prehospital cardiac arrest. Eur J Emerg Med. 2021 Jun 1;28(3):227-232. doi: 10.1097/MEJ.0000000000000786. PMID 33709992
- [Background] Bujak K, Nadolny K, Trzeciak P, Galazkowski R, Ladny JR, Gasior M. Does the presence of physician-staffed emergency medical services improve the prognosis in out-of-hospital cardiac arrest? A propensity score matching analysis. Kardiol Pol. 2022;80(6):685-692. doi: 10.33963/KP.a2022.0109. Epub 2022 Apr 21. PMID 35445741
- [Background] Kern M, Jansen G, Strickmann B, Kerner T. Advancements in Public First Responder Programs for Out-of-Hospital Cardiac Arrest: An Updated Literature Review. Rev Cardiovasc Med. 2025 Jan 22;26(1):26140. doi: 10.31083/RCM26140. eCollection 2025 Jan. PMID 39867188
- [Background] Schwaiger D, Krosbacher A, Eckhardt C, Schausberger L, Baubin M, Rajsic S. Out-of-hospital cardiac arrest: A 10-year analysis of survival and neurological outcomes. Heart Lung. 2025 Sep-Oct;73:1-8. doi: 10.1016/j.hrtlng.2025.04.003. Epub 2025 Apr 18. PMID 40250261
- [Background] Oosterveer DM, de Visser M, Heringhaus C. Improved ROSC rates in out-of-hospital cardiac arrest patients after introduction of a text message alert system for trained volunteers. Neth Heart J. 2023 Jan;31(1):36-41. doi: 10.1007/s12471-021-01656-6. Epub 2022 Jan 6. PMID 34993887
- [Background] Oving I, de Graaf C, Masterson S, Koster RW, Zwinderman AH, Stieglis R, AliHodzic H, Baldi E, Betz S, Cimpoesu D, Folke F, Rupp D, Semeraro F, Truhlar A, Tan HL, Blom MT; ESCAPE-NET Investigators. European first responder systems and differences in return of spontaneous circulation and survival after out-of-hospital cardiac arrest: A study of registry cohorts. Lancet Reg Health Eur. 2020 Nov 20;1:100004. doi: 10.1016/j.lanepe.2020.100004. eCollection 2021 Feb. PMID 35104306
- [Background] Nehme Z, Andrew E, Bernard S, Haskins B, Smith K. Trends in survival from out-of-hospital cardiac arrests defibrillated by paramedics, first responders and bystanders. Resuscitation. 2019 Oct;143:85-91. doi: 10.1016/j.resuscitation.2019.08.018. Epub 2019 Aug 17. PMID 31430512
- [Background] Krammel M, Lobmeyr E, Sulzgruber P, Winnisch M, Weidenauer D, Poppe M, Datler P, Zeiner S, Keferboeck M, Eichelter J, Hamp T, Uray T, Schnaubelt S, Nuernberger A. The impact of a high-quality basic life support police-based first responder system on outcome after out-of-hospital cardiac arrest. PLoS One. 2020 Jun 2;15(6):e0233966. doi: 10.1371/journal.pone.0233966. eCollection 2020. PMID 32484818
- [Background] Siman-Tov M, Strugo R, Podolsky T, Rosenblat I, Blushtein O. Impact of dispatcher assisted CPR on ROSC rates: A National Cohort Study. Am J Emerg Med. 2021 Jun;44:333-338. doi: 10.1016/j.ajem.2020.04.037. Epub 2020 Apr 15. PMID 32336582
- [Background] Salhi RA, Hammond S, Lehrich JL, O'leary M, Kamdar N, Brent C, Mendes de Leon CF, Mendel P, Nelson C, Forbush B, Neumar R, Nallamothu BK, Abir M; CARES Surveillance Group. The association of fire or police first responder initiated interventions with out of hospital cardiac arrest survival. Resuscitation. 2022 May;174:9-15. doi: 10.1016/j.resuscitation.2022.02.026. Epub 2022 Mar 4. PMID 35257834